CLINICAL TRIAL: NCT02693171
Title: A Post-Marketing Study to Further Assess the Immunogenicity and Safety of Unituxin® in High-Risk Neuroblastoma Patients
Brief Title: Post-Marketing Assessment of Immunogenicity and Safety of Unituxin® in High-Risk Neuroblastoma Patients
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: DIV-NB-401
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dinutuximab administered for 5 cycles: High-risk neuroblastoma patient treated with Unituxin as standard of care
  Interventions: Drug: Dinutuximab

INTERVENTIONS:
Drug: Dinutuximab — Unituxin was administered along with cytokines according to the prescribing information
  Other Names: Unituxin®

SUMMARY:
The purpose of this study was to assess the incidence of human anti-chimeric antibody (HACA) in high-risk neuroblastoma patients treated with Unituxin combination therapy.

DETAILED DESCRIPTION:
This was a multi-center, non-randomized, open-label study in patients with high-risk neuroblastoma to assess the immunogenicity, safety and tolerability of Unituxin combination therapy. Patients enrolled in the study were prescribed Unituxin for the treatment of high-risk neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient had been diagnosed with high-risk neuroblastoma.
* Patient had been prescribed Unituxin and plans to start Unituxin therapy within 30 days of study entry.
* Patient started Unituxin therapy no later than 200 days after Autologous Stem Cell Transplantation (ASCT).
* Written informed consent / assent was obtained in accordance with institutional and International Conference on Harmonisation (ICH) guidelines.

Exclusion Criteria:

* Patient had received prior anti-disialoganglioside (anti-GD2) antibody therapy.
* Patient had participated in an investigational clinical trial with tumor therapeutic intent within 30 days of informed consent.
* Patient underwent Autologous Stem Cell Transplantation (ASCT) more than 200 days prior to receiving Unituxin therapy.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High-risk neuroblastoma patients prescribed Unituxin
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ami Desai, MD, Study Chair — Children's Hospital of Philadelphia
Locations (18):
- United States (18):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital- San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center / Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dinutuximab Administered for 5 Cycles
Started | 12 (At study termination, 13 subjects had enrolled, 12 subjects received at least 1 dose of study drug.)
Completed | 3
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Discontinuation of Study by Sponsor | 8

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Dinutuximab Administered for 5 Cycles
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Enrollment
  years | 2.3 (1.37)
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Diagnosis | 1.9 (1.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12
Time since Diagnosis [Mean (Standard Deviation); unit: years] | 0.8 (0.62)
Treatment of Neuroblastoma [Count of Participants; unit: Participants]
  Induction chemotherapy treatment | 12
  Cancer-related surgery | 10
  Single stem cell transplant | 3
  Tandem stem cell transplant | 9
  Radiotherapy treatment | 11
  Other cancer-related treatment | 1
Pre-Autologous Stem Cell Transplantation (ASCT) Response [Count of Participants; unit: Participants]
  Complete response (CR) | 3
  Very good partial response (VGPR) | 6
  Partial response (PR) | 3
  Mixed response (MR) | 0
  No response (NR) | 0
  Progressive disease (PD) | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Incidence of Human Anti-chimeric Antibody (HACA) in High-risk Neuroblastoma Patients Treated With Unituxin Combination Therapy.
Description: Seven blood samples were collected at the following time points for the evaluation of HACA levels:
  * Course 1- Prior to the first Unituxin infusion
  * Course 2- Prior to the first Unituxin infusion
  * Course 3- Prior to the first Unituxin infusion
  * Course 4- Prior to the first Unituxin infusion
  * Course 5- Prior to the first Unituxin infusion
  * Course 6- Prior to the first dose of 13-cis-retinoic acid (RA)
  * Study termination (approximately 2 weeks following the final 13-cis-retinoic acid dose)
Time Frame: Approximately 6 months
Population: Outcome measure data were not collected. Sponsor was required to run this Phase 4 study for EU marketing approval. However, Sponsor terminated the study 15 Dec 2016 and application withdrawn (accepted by European Commission 20 Mar 2017).
Groups:
- Dinutuximab Administered for 5 Cycles: High-risk neuroblastoma patient treated with Unituxin as standard of care
  Dinutuximab: Unituxin will be administered along with cytokines according to the prescribing information
Arm/Group | Dinutuximab Administered for 5 Cycles
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Incidence of Targeted Immune-related Adverse Events (AEs) During Treatment With Dinutuximab Combination Therapy in High-risk Neuroblastoma Subjects.
Description: The incidence of targeted immune-related adverse events (AEs) during treatment with dinutuximab combination therapy in high-risk neuroblastoma subjects were summarized and listed.
Time Frame: Approximately 6 months
Population: Outcome measure data were not collected. Safety data from the 12 subjects dosed prior to study termination were collected and summary level data were reported (eg, total number of subjects affected and total number of events for dinutuximab-treated subjects). Please refer to the adverse event tables for results.
Arm/Group | Dinutuximab Administered for 5 Cycles
Number analyzed (Participants) | 0

3. Secondary Outcome: To Determine the Incidence of Neutralizing Antibody (NAb) in Patients With Human Anti-chimeric Antibody (HACA) Positive Samples.
Description: Incidence of neutralizing antibody (NAb) in patients with human anti-chimeric antibody (HACA) positive samples was summarized and listed.
Time Frame: Approximately 6 months
Population: as for outcome 1
Arm/Group | Dinutuximab Administered for 5 Cycles
Number analyzed (Participants) | 0

4. Secondary Outcome: To Determine the Effect of HACA on Dinutuximab Plasma Concentrations.
Description: Ten blood samples were collected at the following time points for the evaluation of dinutuximab plasma concentrations:
  * Course 1- Prior to the first Unituxin infusion
  * Course 2- Prior to the first Unituxin infusion
  * Course 3- Prior to the first Unituxin infusion
  * Course 4- Prior to the first Unituxin infusion
  * Course 5- Prior to the first Unituxin infusion
  * Course 6- Prior to the first dose of 13-cis-retinoic acid (RA)
  * Study termination (approximately 2 weeks following the final 13-cis-retinoic acid dose).
  An additional 3 blood samples were obtained for the evaluation of dinutuximab plasma concentrations. Each of these blood samples was obtained immediately following the fourth dinutuximab infusion in Courses 1, 3, and 5.
Time Frame: Approximately 6 months
Population: as for outcome 1
Arm/Group | Dinutuximab Administered for 5 Cycles
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The Treatment Phase of the study lasted on average approximately 180 days. From Screening until the completion of study termination assessments, subjects participated in the study for approximately 220 days. However, the Sponsor terminated Study DIV-NB-401 on 15 December 2016; all safety data were collected for each subject from screening until the subject's last scheduled visit.
Arm/Group | Dinutuximab Administered for 5 Cycles
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dinutuximab Administered for 5 Cycles (N=12)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (10)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (8)
Drug eruption (Skin and subcutaneous tissue disorders) | 4 (4)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 8 (15)
Pyrexia (General disorders) | 8 (20)
Adverse drug reaction (General disorders) | 1 (2)
Face oedema (General disorders) | 1 (4)
Oedema (General disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 6 (10)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (15)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Mydriasis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.